CLINICAL TRIAL: NCT07403578
Title: Effect Of Cryotherapy On Anesthetıc Success And Intraoperatıve Paın In Mandıbular Premolars Wıth Irreversıble Pulpıtıs: A Prospectıve Randomızed Clınıcal Trıal
Brief Title: Effect of Cryotherapy on Anesthetic Success and Pain in Irreversible Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayşe Tuğba Eminsoy Avcı, Lecturer, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2026-01-14; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Irreversible Pulpitis; Cryotherapy
MeSH Terms: interventions — Anesthesia, Local; Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- infiltration anesthesia (Experimental)
  Interventions: Procedure: infiltration anesthesia alone; Procedure: infiltration anesthesia combined with cryotherapy
- mandibular anesthesia (Experimental)
  Interventions: Procedure: mandibular anesthesia alone; Procedure: mandibular anesthesia combined with cryotherapy

INTERVENTIONS:
Procedure: infiltration anesthesia alone — Local anesthesia was achieved using buccal infiltration with 2% lidocaine and 1:100,000 epinephrine.
  Arms: infiltration anesthesia
Procedure: mandibular anesthesia alone — Local anesthesia was achieved using mandibular block anesthesia with 2% lidocaine and 1:100,000 epinephrine.
  Arms: mandibular anesthesia
Procedure: infiltration anesthesia combined with cryotherapy — Cryotherapy was applied immediately after completion of the anesthetic injection. Small ice packs wrapped in sterile gauze were placed intraorally on the buccal vestibular surface adjacent to the treated mandibular premolar. Patients were instructed to keep the ice pack in position for 5 minutes. In cases where extreme cold sensation or burning discomfort was reported, patients were asked to remove the ice pack for 1 minute before reapplication
  Arms: infiltration anesthesia
Procedure: mandibular anesthesia combined with cryotherapy — Cryotherapy was applied immediately after completion of the anesthetic injection. Small ice packs wrapped in sterile gauze were placed intraorally on the buccal vestibular surface adjacent to the treated mandibular premolar. Patients were instructed to keep the ice pack in position for 5 minutes. In cases where extreme cold sensation or burning discomfort was reported, patients were asked to remove the ice pack for 1 minute before reapplication
  Arms: mandibular anesthesia

SUMMARY:
This prospective randomized clinical trial aimed to evaluate the effects of different anesthesia protocols on anesthetic success and intraoperative pain during root canal treatment of mandibular premolars diagnosed with symptomatic irreversible pulpitis. A total of 100 systemically healthy patients were randomly allocated into four groups: infiltration anesthesia alone, inferior alveolar nerve block (IANB) alone, infiltration anesthesia combined with cryotherapy, and IANB combined with cryotherapy. Cryotherapy was applied intraorally for 5 minutes immediately after anesthetic administration.

The effectiveness of anesthesia was confirmed using electric pulp testing and cold testing prior to treatment. Root canal therapy was completed in a single visit by a calibrated operator. Intraoperative pain was assessed during access cavity preparation using a visual analogue scale (VAS). Anesthetic success was defined as the presence of no or mild pain, whereas moderate or severe pain indicated anesthetic failure and required supplemental anesthesia.

The primary objective of the study was to determine whether the adjunctive use of cryotherapy improves anesthetic success and reduces intraoperative pain in mandibular premolars with symptomatic irreversible pulpitis. The null hypothesis was that no significant differences would be observed among the study groups in terms of anesthetic success or intraoperative pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients classified as ASA I or II, aged between 18 and 60 years,
* Presence of a restorable mandibular premolar tooth diagnosed with symptomatic irreversible pulpitis,
* History of spontaneous pain or lingering pain elicited by thermal stimuli,
* Positive response with lingering pain to cold testing (Endo Ice; Coltene, Altstätten, Switzerland),
* Positive response at low current levels to electric pulp testing (Parkell Inc., USA),
* Teeth with closed apex and no radiographic evidence of periapical pathology (intact periodontal ligament space and absence of periapical radiolucency),
* Patients presenting with moderate or severe preoperative pain, as assessed using the visual analogue scale (VAS).

Exclusion Criteria:

* Patients who had taken analgesic, anti-inflammatory, or opioid medication within the last 12 hours before treatment,
* Patients with systemic conditions that may affect pain perception, inflammatory response, or healing,
* History of antibiotic use within the previous month or requirement for antibiotic prophylaxis,
* Teeth presenting with clinical or radiographic signs of pulp necrosis or apical periodontitis (Pain on percussion or palpation, presence of sinus tract or swelling, presence of periapical radiolucency),
* Teeth with root resorption, immature apices, severe coronal destruction preventing proper isolation, or calcified canals,
* Teeth that had undergone previous endodontic treatment, including pulpotomy or root canal filling,
* Patients with neurological or psychiatric conditions that could interfere with pain perception or accurate pain reporting,
* Inability to achieve adequate isolation with a rubberdam.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative pain | Baseline/During the Operation
  Intraoperative pain intensity assessed using a Visual Analogue Scale (VAS) (1-10) during access cavity preparation.

IPD SHARING:
Plan to Share IPD: No